CLINICAL TRIAL: NCT05102266
Title: A Randomized, Open-label, Single Dose, Two-way Crossover Phase 1 Study to Evaluate the Pharmacokinetics and Safety of "BR1016C" With "BR1016D" in Healthy Volunteers
Brief Title: A Clinical Trial to Compare the Pharmacokinetics and Safety of "BR1016C" With "BR1016D" in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-SVMC-CT-102
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A(RT) (Experimental): Reference drug "BR1016D" 1 tablet is administered once in fasted state. After having a break of 7 days or more, study drug "BR1016C" 1 tablet is administered once in fasted state.
  Interventions: Drug: BR1016C; Drug: BR1016D
- B(TR) (Experimental): Study drug "BR1016C" 1 tablet is administered once in fasted state. After having a break of 7 days or more, reference drug "BR1016D" 1 tablet is administered once in fasted state.
  Interventions: Drug: BR1016C; Drug: BR1016D

INTERVENTIONS:
Drug: BR1016C — All subjects who have been fasting for at least 10 hours prior to administration will take 1 tablet of study drug or comparator orally with 150 mL of water at room temperature at around 8 a.m. on the administration day of each period.
  Other Names: Study drug
Drug: BR1016D — All subjects who have been fasting for at least 10 hours prior to administration will take 1 tablet of study drug or comparator orally with 150 mL of water at room temperature at around 8 a.m. on the administration day of each period.
  Other Names: Reference drug

SUMMARY:
To evaluate the pharmacokinetic properties and safety of "BR1016C" and "BR1016D" in healthy adults.

DETAILED DESCRIPTION:
Descriptive statistics (number of subjects, mean, standard deviation, median, minimum, maximum, etc.) will be presented for continuous data, and the number (N) and percentage (%) of subjects for each category will be summarized and presented for categorical data. For pharmacokinetic data, the number of subjects, mean, standard deviation, coefficient of variation (primary endpoint only), median, minimum, and maximum will be presented by treatment group.

<Demographic information statistical analysis>

* Descriptive statistical analysis will be performed on basic data including demographic information (gender, age, height, weight, BMI, etc.) of all randomized subjects (Intention-To-Treat).
* Continuous data will be compared and tested between sequence groups by summarizing descriptive statistics (number of subjects, mean, standard deviation, median, minimum, maximum, etc.), and by testing whether the data are normally distributed using the independent t-test or Wilcoxon's rank sum test. For categorical data, the number (N) and percentage (%) of subjects for each category will be summarized and compared between the order groups using a Chi-square test or Fisher's exact test.

<Pharmacokinetic statistical analysis>

* The pharmacokinetic assessment will be analyzed in subjects who can complete all scheduled blood sampling for pharmacokinetic assessment after administration of the investigational product according to the protocol and can be assessed for pharmacokinetics, and there are no major protocol violations that may affect the pharmacokinetic analysis.
* The pharmacokinetic assessment will be conducted in accordance with Article 17 of the "Drug Equivalence Test Criteria" and the pharmacokinetic parameters will be calculated using a noncompartmental method using the software 'Phoenix® Winnonlin® Ver.8.3 (or higher) (Certara L.P.)'. When calculating pharmacokinetic parameters, the actual sampling time will be used for the sampling time for each subject, and the linear trapezoidal method will be used for the calculation of AUCt. Pharmacokinetic parameters will be summarized and presented descriptively by subject and treatment group. For statistical analysis for equivalence assessment, analysis of variance will be performed for log-transformed values of AUCt and Cmax at a significance level of 0.05. If the 90% confidence interval of the difference between the control drug and the mean value of the study drug is within log 0.8 to log 1.25, the control drug and the study drug will be assessed as equivalent. Descriptive statistics will be presented by treatment group, and they will be compared between treatment groups if necessary.
* The analysis of variance will test the administration period (period), sequence group (sequence), and treatment group (treatment) as fixed effects, and the difference between individuals as linear mixed effect model considering random effects.

<Safety statistical analysis>

* The analysis set for safety assessment includes all subjects who received the investigational product at least once.
* Adverse events will be assessed based on the treatment-emergent adverse events (TEAEs) that occur after the administration of the investigational product in Period 1. For TEAEs that occurred during the washout period, hospital admission date, and prior to administration, it will be determined as a TEAE of the investigational product that was administered previously.

Adverse event names will be standardized by SOC (System Organ Class) and PT (Preferred Term) terms using the MedDRA (version 24.0 or higher) classification system, and the analysis of adverse events will be presented as the number of subjects who experienced adverse events, incidence (%), and number of occurrences based on TEAEs. The severity, seriousness, and causal relationship to the investigational product of adverse events will be summarized by treatment group. If necessary, the Chi-square test, Fisher's exact test or McNemar's test will be conducted to test for inter-group differences.

* The names of concomitant medications will be standardized using the WHO ATC (2021 or later) classification system, and subjects who received concomitant medications during the clinical study will be listed. In case of concomitant medications taken during the washout period, hospital admission date, or before the administration, it shall be determined as the concomitant medication of the investigational product that was administered previously.
* For other observation and test items of the subjects such as clinical laboratory tests, vital signs, electrocardiography (ECG), and physical examinations, descriptive statistical analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 19 years or older at screening
2. Individuals with an index BMI of 18.0 to 30.0 for obesity (BMI calculation: weight (kg)/height (m)2)

   * Males weighing 50 kg or more
   * Females weighing 45 kg or more
3. Those who do not have clinically significant congenital or chronic diseases and do not have pathological symptoms or findings as a result of medical examination (electroencephalography, electrocardiogram, chest and stomach endoscopy or gastrointestinal radiography, if necessary)
4. A person who has been determined by the principal investigator (or a delegated sub-investigator) to be eligible as a subject based on the results of electrocardiography (ECG) and clinical laboratory tests such as hematology, blood chemistry, serology, urinalysis, etc. conducted according to the properties of the drug
5. Those who voluntarily decided to participate in the study after being given a detailed explanation of this clinical trial and understanding it fully, and provided a written consent to follow the precautions during the clinical study period
6. Those who agreed to rule out the possibility of a pregnancy by using a medically accepted method of contraception* for themselves, their spouse, or their partner from the date of screening until 7 days after the date of the last investigational product administration and agreed not to provide sperm or eggs *Medically acceptable methods of contraception: Combined use of intrauterine device (IUD, IUS), vasectomy, tubal ligation and barrier methods (male condom, female condom, cervical cap, diaphragm, sponge, etc.) or combined use of two or more barrier methods if spermicide is used

Exclusion Criteria:

1. Those who have taken drugs that induce and inhibit drug metabolizing enzymes such as barbitals within 30 days prior to the initiation of the study (date of first administration) or who have taken drugs that may interfere with this study within 10 days prior to the initiation of the study (date of first administration)
2. Those who have participated in a bioequivalence study or other clinical study within 180 days prior to the initiation of the study (date of first administration) and have received the investigational product
3. Those who have donated whole blood or blood within 60 days prior to the first day of administration, or donated blood components within 14 days prior to the first day of administration or who have received a blood transfusion within 30 days
4. Those who have gastrointestinal disease or history of gastrointestinal resection (except for hernia surgery or simple appendectomy) that may affect the absorption of the drug
5. Those who have continued drinking alcohol within 30 days prior to the initiation of the study (date of first administration)

   * Male: 4 drinks/time, more than 14 drinks/week
   * Female: 3 drinks/time, more than 7 drinks/week (1 drink: 45 mL of spirits, 150 mL of wine, 350-360 mL of beer, 300 mL of makgeolli, 90 mL of 20% soju)
6. Smokers who smoked more than 10 cigarettes a day within the 90 days prior to the initiation of the study (date of first administration) and who are unable to stop smoking from 48 hours prior to the first administration of the investigational product until the last blood collection
7. Those who have ingested or cannot refrain from ingesting caffeine-containing foods (e.g., coffee, green tea, tea, soda, coffee milk, sour tonic drinks, etc.) from 48 hours prior to the initiation of the study (date of first administration) until the last blood collection
8. Those who have had an abnormal diet that may affect the absorption, distribution, metabolism, and excretion of the drug (e.g., consumption of grapefruit juice (at least 1L per day) within 7 days prior to administration of the investigational product)
9. Those who meet any of the criteria below in the clinical laboratory test results at screening

   * AST (SGOT) or ALT (SGPT) or γ-GTP levels in blood greater than 1.5 times the upper limit of the normal range (ULN)
   * eGFR < 60mL/min/1.73 m2
   * Sodium(Na) < 135 mEq/l
   * Potassium(K) > 5.0 mEq/l
   * Positive results in HBsAg, HCV-Ab, HIV antibody, and VDRL (Syphilis/qualitative) test
10. Those who meet any of the criteria below in the results of vital sign measurement at screening

    * Systolic blood pressure: Less than 90 mmHg or more than 139 mmHg
    * Diastolic blood pressure: Less than 60 mmHg or more than 90 mmHg
    * Pulse rate: Greater than 100/min
11. Patients with the following conditions

    * Those who have a hypersensitivity reaction to the active ingredient of this drug or to any component of this drug
    * Those who are receiving an angiotensin-converting enzyme (ACE) inhibitor or have not passed 36 hours after discontinuing the administration
    * Those who have a history of angioedema when angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor antagonist (ARB) was administered
    * Those with hereditary or idiopathic angioedema
    * Severe hepatic impairment, cirrhosis or biliary obstruction, cholestasis
    * Those who are receiving a combination administration with aliskiren for diabetes or moderate to severe renal impairment (eGFR < 60mL/min/1.73 m2)
    * Those with primary hyperaldosteronism
12. Those with a history of clinically significant psychiatric illness within 5 years prior to the screening visit
13. For female volunteers, pregnant women or those who may be pregnant or are breastfeeding
14. Individuals who the principal investigator (or a delegated sub-investigator) has determined to be ineligible for this clinical study for reasons other than the inclusion/exclusion criteria described above

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
AUCt of BR1016C and BR1016D | 0-36 hours after administration
  Area under the plasma drug concentration-time curve of BR1016C and BR1016D
Cmax of BR1016C and BR1016D | 0-36 hours after administration
  Maximum concentration of drug in plasma of BR1016C and BR1016D

SECONDARY OUTCOMES:
AUC∞, AUCt/AUC∞, Tmax, t1/2, CL/F and Vz/F of BR1016C and BR1016D | 0-36 hours after administration
  AUC∞, AUCt/AUC∞, Tmax, t1/2, CL/F and Vz/F of BR1016C and BR1016D

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Min Seong, Principal Investigator — Bestian Hospital
Locations (1):
- Bestian Hospital, Osŏng, South Korea

IPD SHARING:
Plan to Share IPD: No